CLINICAL TRIAL: NCT00846391
Title: A Phase IIa, Multicenter, Double-Blind, Placebo-Controlled Clinical Trial to Study the Efficacy and Safety of MK8245 in Patients With Type 2 Diabetes Mellitus With Inadequate Glycemic Control
Brief Title: A Study to Assess the Safety and Efficacy of MK8245 in Patients With Type 2 Diabetes Mellitus and Inadequate Glycemic Control (MK8245-005 AM2)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to inability to recruit patients.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8245-005; 2009_541
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2010-09-21 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (5-(3-(4-(2-bromo-5-fluorophenoxy)piperidin-1-yl)isoxazol-5-yl)-2H-tetrazol-2-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MK8245 5 mg b.i.d. (Experimental): MK8245
  Interventions: Drug: MK8245 5 mg (twice a day) b.i.d.
- MK8245 50 mg b.i.d. (Experimental): MK8245
  Interventions: Drug: MK8245 50 mg b.i.d.
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK8245 5 mg (twice a day) b.i.d. — All patients will receive placebo capsules 2 weeks prior to treatment period to be taken twice daily.
  Patients randomized to the 5 mg b.i.d. treatment group took 2 capsules of MK8245 2.5 mg in the morning and 2 capsules of MK8245 2.5 mg in the evening.
  Other Names: MK8245
  Arms: MK8245 5 mg b.i.d.
Drug: MK8245 50 mg b.i.d. — All patients will receive placebo capsules 2 weeks prior to treatment period to be taken twice daily.
  Patients randomized to the 50 mg b.i.d. treatment group took 2 capsules of MK8245 25 mg in the morning and 2 capsules of MK8245 25 mg in the evening.
  Other Names: MK8245
  Arms: MK8245 50 mg b.i.d.
Drug: Placebo — All patients will receive placebo capsules 2 weeks prior to treatment period to be taken twice daily.
  Patients randomized to the placebo treatment group took 2 capsules of placebo matching MK8245 capsules in the morning and 2 placebo capsules matching MK8245 capsules in the evening.
  Arms: Placebo

SUMMARY:
A study to assess the safety and efficacy of MK8245 as monotherapy compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes Mellitus
* 18 to 65 years of age

Exclusion Criteria:

* History of Type 1 Diabetes or ketoacidosis
* Have been treated with lipid lowering medications 4 weeks before starting the study
* Have started on a weight loss program and not in the maintenance phase or have started weight loss medication within the last 12 weeks
* Have had surgery in the last 30 days
* History of active liver disease
* History of coronary heart disease or congestive heart failure
* Have had a stroke or transient ischemic neurological disorder in the past 6 months
* Are Human Immunodeficiency Virus (HIV) Positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In:10-Feb-2009
  Early Termination*:11-Aug-2009
  Last Patient Last Visit:19-Aug-2009
  10 Centers Worldwide
  *Study was terminated due to inability to recruit patients. Because it was not terminated for safety concerns, sites were to see patients for early termination visit at earliest convenience. The last patient was seen 19-Aug-2009.
Pre-assignment Details: Patients 18-65 yrs not on antihyperglycemic agent (AHA) (A1C 7-10%),or single AHA (A1C 7-9.5%),or low dose dual AHA therapy (A1C 6.5-9.5%) with type 2 diabetes mellitus entered a 4-wk diet/exercise period (AHA wash-off if on AHA),after which,those with fasting glucose of 130-250 mg/dL were eligible for randomization (after a 2 wk pbo run-in period)
Groups:
- MK8245 5 mg b.i.d.: Patients randomized to the 5 mg (twice a day) b.i.d. treatment group took 2 capsules of MK8245 2.5 mg in the morning and 2 capsules of MK8245 2.5 mg in the evening.
- MK8245 50 mg b.i.d.: Patients randomized to the 50 mg b.i.d. treatment group took 2 capsules of MK8245 25 mg in the morning and 2 capsules of MK8245 25 mg in the evening.
- Placebo: Patients randomized to the placebo treatment group took 2 capsules of placebo matching MK8245 capsules in the morning and 2 placebo capsules matching MK8245 capsules in the evening.
Period: Overall Study
Arm/Group | MK8245 5 mg b.i.d. | MK8245 50 mg b.i.d. | Placebo
Started | 4 | 4 | 6
Completed | 3 | 2 | 3
Not Completed | 1 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK8245 5 mg b.i.d. | MK8245 50 mg b.i.d. | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (13.4) | 55.5 (7.7) | 53.5 (7.5) | 53.0 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 2 | 0 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 2 | 2 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black OR African American | 0 | 0 | 1 | 1
  Multi-Racial | 1 | 0 | 0 | 1
  White | 3 | 4 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 24-hour Weighted Mean Glucose (WMG) at Week 4
Description: The 24-hour WMG is derived from multiple glucose values collected during both fasting and post-meal periods. A "weighted" rather than a "simple" mean is used to avoid overrepresentation of post-meal glucose values.
  Blood samples for glucose were to be collected immediately prior to (sample -10 minutes), and 0, 15, 30, 60, 90, 120, and 180 minutes after each meal, and overnight (at midnight, 3 AM, and 5 AM) and fasting at 7 AM. Patients were to be domiciled for approximately 26 hours at the site where standard meals were provided and physical activity monitored.
Time Frame: Baseline and Week 4
Population: The analysis population included all patients with a baseline value and Week 4 value for this outcome.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MK8245 5 mg b.i.d. | MK8245 50 mg b.i.d. | Placebo
Number analyzed (Participants) | 3 | 2 | 3
mg/dL | -18.9 (22.1) | 18.7 (6.7) | -12.6 (1.4)

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from Visit 2 (Week -6) through Visit 6 (Week 4). Serious adverse experiences were collected for up to 14 days after the last dose of study medication.
Arm/Group | MK8245 5 mg b.i.d. | MK8245 50 mg b.i.d. | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 3/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK8245 5 mg b.i.d. (N=4) | MK8245 50 mg b.i.d. (N=4) | Placebo (N=6)
Punctate keratitis (Eye disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headadache (Nervous system disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
This study was terminated due to the continuing inability to recruit patients. No efficacy analysis was performed because of insufficient sample size for meaningful analysis due to early study termination and insufficient sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.